CLINICAL TRIAL: NCT04149652
Title: Role of Lung Ultrasonography for Detecting COPD and Fibrosis and Stratifying the Risk of COPD in Healthy Subjects
Brief Title: Lung Elastrosonography in Diagnosis and Stratification of COPD and Fibrosis
Acronym: ELAS-P-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Tiziana Meschi, Head of Geriatric-Rehabilitation Department, Associate Professor of Internal Medicine, Azienda Ospedaliero-Universitaria di Parma
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 614/2018/DISP/AOUPR
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Smoker Lung
Keywords: elastography; ultrasound; copd; smoke; lung stiffness; lung ultrasound
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Experimental study of feasibility of an ultrasound technique for diagnostic purposes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with COPD or fibrosis (Other): Subjects, enrolled on either an inpatient or outpatient basis, with stable COPD or fibrosis documented by anamnestic, imaging and functional tests. They will undergo lung function tests and bedside lung ultrasound integrated with lung elastosonography.
  Interventions: Diagnostic Test: Lung Elastosonography
- Smokers with no signs of COPD (Other): Subjects with an active smoking habit or a personal history of hard smoking dating back to maximum 5 years before, without clinical and functional signs of COPD. They will undergo lung function tests and bedside lung ultrasound integrated with lung elastosonography.
  Interventions: Diagnostic Test: Lung Elastosonography
- Healthy non-smoking volunteers (Other): Healthy volunteers who have never smoked and who have no clinical or functional sign of COPD or other respiratory diseases. They will undergo lung function tests and bedside lung ultrasound integrated with lung elastosonography.
  Interventions: Diagnostic Test: Lung Elastosonography

INTERVENTIONS:
Diagnostic Test: Lung Elastosonography — Bedside lung ultrasound integrated with lung elastosonography, performed by using the convex probe of an Esaote Mylab Seven ultrasound system (Esaote, Genova, Italy), equipped with the strain elastography module ElaXto©.
  Other Names: Lung Elastography

SUMMARY:
Elastosonography is an advanced ultrasound technique, nowadays available in many portable systems, allowing to measure elasticity and stiffness of parenchymatous organs. Its main current applications concern the advanced diagnostics of liver, thyroid and breast nodules. Few studies have applied elastosonography to the respiratory system, and to date no-one has evaluated the elasticity of lung parenchyma in COPD and only one in pulmonary fibrosis. The primary aim of this study is to compare the elasticity features of lung parenchyma, measured by bedside ultrasound integrated with ultrasonography, among three groups of subjects: 1. patients with COPD and/or lung fibrosis; 2. smokers with no functional evidence of COPD or fibrosis; 3. healthy non-smoking volunteers. The secondary aim is to verify the possible correlation of elastosonography-related parameters of lung elasticity/stiffness with results of lung function tests.

One hundred and thirty-eight subjects (46 per group) will be enrolled in this experimental study, on both inpatient and outpatient basis. The presence or absence of COPD or fibrosis will be assessed integrating personal history, imaging tests and functional tests prior to enrolment. Smoking habits will also be carefully investigated. Excluded from the study will be all subjects with acute COPD flares, acute respiratory failure, inability to undergo lung ultrasound examination and lung function tests, cognitive impairment, severe motoric disability, cancer, poor survival prognosis.

Each participant will undergo standard lung function tests and bediside ultrasound examination integrated with lung elastosonography during the same day. Lung function tests will be performed with a Carefusion MSC Body spirometer following standard procedures. Lung ultrasound will be performed by a skilled physician, using the convex probe of an Esaote Mylab Seven ultrasound system (Esaote, Genova, Italy), equipped with strain elastography module ElaXto©. The participant will remain in the sitting position for the whole ultrasound/elastography procedure, with the examiner systematically scanning intercostal spaces on both sides of the back thorax. After performing a standard lung ultrasound scan to verify the absence of consolidations or signs of respiratory diseases other than COPD, the examiner will activate the elastography module, performing little compressions with the wrist on the convex probe, to obtain adequate elastography images combining ranges of red, green and blue colors. Images will then be analyzed with the software ElaXto©, to obtain the percentage of stiffness in areas of interest of lung parenchyma.

Statistical analyses will be focused on comparison of stiffness index across different groups, and on correlation of elastosonographic parameters with lung function tests (FEV1, Tiffeneau index).

DETAILED DESCRIPTION:
Introduction

Chronic Obstructive Pulmonary Disease (COPD) is a common respiratory disease characterized by irreversible expiratory airflow limitation with bronchial hyperinflation and air trapping, causing a reduction of pulmonary and thoracic compliance, characterized by chronic inflammation with emphysematous destruction of the lungs (GOLD Guidelines 2019; Singh P et al 2019; Bagdonas E et al 2015).

In the last decade, bedside lung ultrasonography (LUS) has rapidly gained popularity for the differential diagnosis of respiratory diseases, especially in the acute setting, for its accuracy, repeatability, rapidity and versatility that make it the ideal diagnostic tool in the internal medicine and geriatric setting (Ticinesi A et al 2019).

COPD is not associated with any specific sign at LUS, so that, in a context of acute exacerbation with respiratory failure, it remains a diagnosis of exclusion (Lichtenstein D 2015). Instead, lung function tests (i.e., spirometry) is considered the gold standard test for COPD detection (GOLD Guidelines 2019).

However, spirometry suffers from some limits, the major being its dependence on the cooperation of the subject, because during the test it is necessary to perform a correct expiratory forced manoeuvre with restricted acceptability standards (American Thoracic Society 1991; American Toracic Society 1995). As such, it can not be perfomed in patients with severe cognitive and physical impairment. Furthermore, spirometry is contraindicated in many conditions which may be aggravated by the effort (i.e. unstable cardiovascular status, recent myocardial infarction, pulmonary embolism and other) (American Association for Respiratory Care 1996). Alternative methods of identification of COPD and stratification of its risk in clinical practice are thus highly desirable, but unavailable to date.

Interstitial lung disease (ILD) represents a wide range of lung pathologies characterized by connective tissue deposition and fibrous remodeling of the lungs, causing a severe and progressive loss of respiratory function (Meyer KC 2017). High-resolution computed tomography (HRCT) is currently considered the gold standard in diagnosing and monitoring ILD, but, in its use, it is necessary to consider the ionizing radiation exposure (the cumulative dose for each exam is estimated around 7mSv, equivalent to two years of sunlight exposure), which may affect the repeatability of the exam, the high cost and the unavailability in many hospitals.

Moreover, because of main alveolar involvement in ILD, LUS can show a variable number of B-lines, even if this is a non-specific artifact common to other pathologic lung conditions (i.e. heart failure with pulmonary oedema and acute respiratory distress syndrome), and a thickening of pleural line greater than 3 mm (Wohlgenannt S et al 2001).

Pathophysiological basis of COPD and ILD allow to assume that lung parenchyma of these patients is stiffer than the normal one, but easy tools for measuring lung parenchyma stiffness in vivo are still lacking in clinical practice.

Elastography is a noninvasive diagnostic tool, complementary to ultrasonography, that assess in real-time the parenchymal elasticity degree, evaluating tissue mechanical properties (Gennisson JL et al 2013). Currently, this technique is widely used to study liver fibrosis and characterize suspect nodules and lesions of breast, thyroid, kidney and prostate (Gennisson JL et al 2013).

At present, only one study (Zhang X et al 2019) has considered the role of surface wave elastography in measuring the elastic properties of superficial lung tissue in patients with ILD, but there are not studies concerning its application in COPD for diagnostic purposes or for stratifying the risk of onset of the disease in smokers.

The aim of this study is to evaluate the applicability of strain elastography, integrated with LUS, in the assessment of the risk and the diagnosis of COPD and ILD.

Study hypothesis

The main hypothesis of the study is that the use of surface wave strain elastography during execution of a chest ultrasound examination is able to differentiate subjects suffering by COPD or ILD and subjects who have not respiratory diseases, documenting different stiffness properties of lungs. Another hypothesis is that the lungs of active smokers or ex-smokers with a long exposure to smoke exhibit a different stiffness pattern than that of the lungs of healthy non-smokers at elastosonographic examinations. Finally, another hyothesis is that the anatomical damage detected by lung ultrasonography is significantly correlated with parameters of lung function tests.

Objectives

1. To compare the stiffness properties of lung parenchyma, measured in vivo by lung ultrasound integrated with surface wave strain elastography, across three different groups of subjects: one group with established diagnosis of COPD or fibrosis, one group with no chronic lung diseases but high risk of developing COPD (i.e., active smokers or ex-smokers), and one group of healthy non-smokers.
2. To verify the possible correlations of stiffness properties of lung parenchyma, as measured by surface wave strain elastography, with lung function tests.

Study design

Single-center experimental diagnostic study, no profit and not involving drugs.

Setting

The study will be performed and completed at the Internal Medicine and Critical Subacute Care Unit of Parma University-Hospital, Italy. The unit is a large internal medicine area (100 beds for inpatients) dedicated to the care of older patients. It also includes an outpatient area where ultrasound and spirometry diagnostic resources are available. Both inpatients and outpatients will be involved in the study.

Study population

One-hundred thirty-eight participants will be enrolled (46 per group). The COPD/fibrosis group must have anamnestic record of chronic respiratory disease (COPD or ILD), confirmed by recent imaging and/or spirometric findings. The "high risk" group must be composed of active smokers or ex-smokers with significant exposure dating back to no more than 5 years and high risk of COPD according to the GOLD Guidelines 2019. The "healthy" group must have never smoked and have no record of chronic respiratory diseases. Excluded will be all subjects with acute respiratory failure not allowing to undergo study procedures, cognitive impairment or dementia, severe mobility disability, severe neuromuscular diseases, severe heart failure, severe kidney or liver disease, cancer or lack of compliance to study procedures (exclusion criteria common to all groups).

The sample size is set at 138 participants (46 per group) basing on a temptative calculation supposing the non-inferiority of lung elastography as compared with spirometry (sensitivity not lower than 10%) in detecting COPD or ILD (alpha=0.05, precision 5%). However, a precise sample size calculation is not possible due to the complete absence of clinical data on the diagnostic relevance of elastography in COPD.

Study procedures

Participants will be enrolled either on an inpatient or outpatient basis, provided that they fulfil all inclusion criteria for the respective group and that they do not have any of the exclusion criteria. The enrolment of volunteers will be also supported by the use of flyers and public notices.

After obtaining written informed consent and consent to personal data management (according to the European Union GDPR Regulation 2016/679), all participants will be evaluated by a staff physician collecting personal history and basic clinical data, if available. Collected data will include age, presence or absence of respiratory diseases (especially COPD and ILD), comorbidities, chronic drug treatments, most recent laboratory tests, reports of most recent chest imaging examinations, reports of most recent lung function tests. Smoking habits will be carefully assessed, with special attention on timing of the habit and quantity of cigarettes.

Lung function tests will be then performed following standard and internationally recognized protocols (American Association for Respiratory Care 1996), by using a Carefusion MSC Body spirometer. FEV1 and Tiffeneau Index (FEV1/FVC) will be particularly assessed.

Lung ultrasound will then be performed by a staff physician, by means of a Esaote Mylab Seven ultrasound system (Esaote, Genova, Italy), equipped with the strain elastography module ElaXto©. The examinations will be all performed using a convex 3.5-5 mHz probe, with the participant in sitting position and the examiner behind him or her.

First, the physician will perform a routine B-mode lung ultrasound, exploring both lungs in order to rule out other diseases which could influence pulmonary and thoracic compliance and lung parenchyma elasticity. Then, the physician will activate the elastography module and performe little compressions on the convex probe with the wrist, according to ultrasound detector, to obtain elastography images suitable for color analysis. Elastography images are in fact composed of a mix of red, green and blue colors, whose combination is an expression of the stiffness of the examined parenchyma. The examiner will perform a systematic bilateral scan, beginning from posterior lung areas, two intercostal spaces above diaphragm, and acquiring two images for each side, a basal one and an apical one. The examiner will then move to lung lateral regions, to the base of safety triangle, acquiring other two images, a basal one and an apical one, and finally to lung anterior regions, at the third intercostal space on the mid-clavicular line on the right side and at the second intercostal space on the mid-clavicular line on the left side (to avoid the cardiac area), acquiring other two images, a basal one and an apical one, for a total of 12 scans per participant.

Elastography images will be archived on ultrasound system and subsequently analysed in post-processing on the specific ultrasound software ElaXto©. Through this software, it is possible to measure qualitatively the percentage of tissue elasticity and stiffness.

For each image, the percentage of stiffness, with a stiffness threshold set at 20%, will measured in three areas of interest, by using the manual trace:

* The total area of lung parenchyma explored (excluding subcutaneous and muscular tissue located above the pleural line);
* The superficial half of lung parenchyma explored area (until approximately 3-4 cm under the pleural line);
* The deep half of lung parenchyma explored area (from 3-4 cm of depth until the lower limit of the image).

The use of three different stiffness measures for each image assures to highlight the overall stiffness of the explored lung parenchyma, as well as potential regional differences between the superficial and the deep lung plans. In fact, COPD is expected to mainly involve deeper portions of lung parenchyma, being basically a disease of small airways, while ILD is expected to mainly involve superficial plans of lung parenchyma (subpleural fibrosis). For each image, a qualitative index of elasticity and a quantitative index of stiffness will be obtained.

All the examinations on participants will be performed during the same day.

Statistical analysis

Data will be expressed as median and interquartile range or mean plus/minus standard deviation, according to variable distribution. Elastography parameters will be compared across the three study groups by means of ANCOVA and Bonferroni test. The correlations between spirometric and elastographic parameters will be assessed by Pearson correlation index.

Ethical issues

Spirometry and elastosonography are two safe examinations not implying any specific risk for participants. All procedures will follow the Good Clinical Practice and Declaration of Helsinki principles. Data will be handled in compliance with the current European Union legislation.

ELIGIBILITY:
Inclusion Criteria:

COPD/fibrosis group

* Established anamnestic record of COPD or fibrosis confirmed by imaging and functional tests
* Capacity to maintain the sitting position for chest ultrasound
* Capacity and willingness to collaborate to the execution of lung function tests

Smoker group

* Active smoking habit or personal history of hard smoking (at least 10 cigarettes/day) in the five year period before evaluation
* Presence of a high risk of COPD according to GOLD guidelines
* No anamnestic, clinical or functional evidence of COPD
* Capacity to maintain the sitting position for chest ultrasound
* Capacity and willingness to collaborate to the execution of lung function tests

Healthy non-smoking volunteer group

* Absence of a current or past smoking habit
* Absence of a high risk of COPD according to GOLD guidelines
* Capacity to maintain the sitting position for chest ultrasound
* Capacity and willingness to collaborate to the execution of lung function tests

Exclusion Criteria:

* Acute respiratory failure
* Cognitive impairment or dementia
* Severe motoric disability with inability to maintain the sitting position
* Lung diseases
* Severe heart failure
* Severe kidney or liver failure
* Cancer
* Severe neuromuscular diseases
* Any other condition that could represent a bias for the accuracy of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Elasticity score of lung parenchyma | The same moment of baseline evaluation
  Qualitative index of elasticity measured by lung ultrasonography (visual score ranging from 1 to 3, 1=elastic pattern 3=rigid pattern)
Strain index of lung parenchyma | The same moment of baseline evaluation
  Quantitative index of stiffness of lung parenchyma measured by lung ultrasonography (percentage of stiffness ranging from 0% to 100%, with 100% representing extreme rigidity)

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Meschi, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma (Parma University Hospital)
Locations (1):
- UO Medicina Interna e Lungodegenza Critica, Azienda Ospedaliero-Universitaria di Parma, Parma, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No
IPD, and especially ultrasound images, will not be made available due to privacy law restrictions. Aggregated data will be made available in anonymous form upon reasonable request.

REFERENCES:
- [Background] Singh D, Agusti A, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Criner GJ, Frith P, Halpin DMG, Han M, Lopez Varela MV, Martinez F, Montes de Oca M, Papi A, Pavord ID, Roche N, Sin DD, Stockley R, Vestbo J, Wedzicha JA, Vogelmeier C. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease: the GOLD science committee report 2019. Eur Respir J. 2019 May 18;53(5):1900164. doi: 10.1183/13993003.00164-2019. Print 2019 May. PMID 30846476
- [Background] Ticinesi A, Scarlata S, Nouvenne A, Lauretani F, Incalzi RA, Ungar A; GRETA (Gruppo di Ricerca sull'Ecografia Toracica nell'Anziano) Group of the Italian Society of Gerontology and Geriatrics (SIGG). The Geriatric Patient: The Ideal One for Chest Ultrasonography? A Review From the Chest Ultrasound in the Elderly Study Group (GRETA) of the Italian Society of Gerontology and Geriatrics (SIGG). J Am Med Dir Assoc. 2020 Apr;21(4):447-454.e6. doi: 10.1016/j.jamda.2019.06.018. Epub 2019 Aug 6. PMID 31399360
- [Background] Lichtenstein DA. BLUE-protocol and FALLS-protocol: two applications of lung ultrasound in the critically ill. Chest. 2015 Jun;147(6):1659-1670. doi: 10.1378/chest.14-1313. PMID 26033127
- [Background] Bagdonas E, Raudoniute J, Bruzauskaite I, Aldonyte R. Novel aspects of pathogenesis and regeneration mechanisms in COPD. Int J Chron Obstruct Pulmon Dis. 2015 Jun 2;10:995-1013. doi: 10.2147/COPD.S82518. eCollection 2015. PMID 26082624
- [Background] Lung function testing: selection of reference values and interpretative strategies. American Thoracic Society. Am Rev Respir Dis. 1991 Nov;144(5):1202-18. doi: 10.1164/ajrccm/144.5.1202. No abstract available. PMID 1952453
- [Background] Standardization of Spirometry, 1994 Update. American Thoracic Society. Am J Respir Crit Care Med. 1995 Sep;152(3):1107-36. doi: 10.1164/ajrccm.152.3.7663792. No abstract available.
- [Background] Meyer KC. Pulmonary fibrosis, part I: epidemiology, pathogenesis, and diagnosis. Expert Rev Respir Med. 2017 May;11(5):343-359. doi: 10.1080/17476348.2017.1312346. Epub 2017 Apr 10. PMID 28345383
- [Background] Wohlgenannt S, Gehmacher O, Gehmacher U, Kopf A, Mathis G. [Sonographic findings in interstitial lung diseases]. Ultraschall Med. 2001 Feb;22(1):27-31. doi: 10.1055/s-2001-11252. German. PMID 11253553
- [Background] Gennisson JL, Deffieux T, Fink M, Tanter M. Ultrasound elastography: principles and techniques. Diagn Interv Imaging. 2013 May;94(5):487-95. doi: 10.1016/j.diii.2013.01.022. Epub 2013 Apr 22. PMID 23619292
- [Background] Zhang X, Osborn T, Zhou B, Meixner D, Kinnick RR, Bartholmai B, Greenleaf JF, Kalra S. Lung Ultrasound Surface Wave Elastography: A Pilot Clinical Study. IEEE Trans Ultrason Ferroelectr Freq Control. 2017 Sep;64(9):1298-1304. doi: 10.1109/TUFFC.2017.2707981. PMID 28866480
- See also: GOLD Guidelines 2019 — https://goldcopd.org/wp-content/uploads/2018/11/GOLD-2019-v1.7-FINAL-14Nov2018-WMS.pdf